CLINICAL TRIAL: NCT02590354
Title: Analytical Treatment Interruption in HIV Positive Patients With Low Viral Reservoir to Evaluate the Potential of a Functional Cure
Brief Title: Analytical Treatment Interruption in HIV Positive Patients
Acronym: ISALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: University Hospital, Ghent (Other); Universitair Ziekenhuis Brussel (Other); Saint-Pierre University Hospital (Other); Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ITM0714
Record Dates: First submitted 2015-10-14; First posted 2015-10-29 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: HIV-1 Infection
Keywords: Treatment interruption; functional cure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment interruption (Experimental): The ART treatment in patients with a very low viral reservoir will be interrupted.
  Interventions: Other: ART interruption

INTERVENTIONS:
Other: ART interruption

SUMMARY:
HIV-1 infected patients with normal peripheral blood CD4+ T-cell counts and undetectable viral load will be recruited in four Belgian HIV reference centers. Selected patients will undergo a two-step screening in which a viral reservoir measurement will be performed and among those with a very low viral reservoir an analytical treatment interruption of their longstanding antiretroviral therapy (ART). There is no randomization foreseen. Patients will receive an intense clinical and laboratory follow-up during 48 weeks followed by 12 weeks post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent
* Men and women age ≥ 18 and < 65 years.
* Confirmed HIV-1 infection at any time prior to study entry.
* Infected with HIV-1 subtype A, B, C, D, CRF01_AE or CRF02_AG virus
* Participant should take ART for at least 2 years before baseline with no changes in the ART regimen for at least 90 days prior to study entry. ART regimen is defined as mono- or bi-therapy or a combination of three or more active antiretroviral drugs
* CD4 T-cell count is >= 500/μl for a period of at least 3 months prior study entry
* Nadir CD4+ T-cell count is ≥300/μl. A lower nadir CD4+ T-cell count will be allowed if measured at time of acute infection as far as the relative CD4+ count remains above 20%. An acute infection is defined as an association of a clinical picture of retroviral syndrome together with a seroconversion in HIV serology or an incomplete confirmation test.
* Plasma viral load < 50 copies/ml for at least 2 years before baseline. (Occasional "blips" will be permitted if it happened more than six months before study entry. An occasional blip is defined as an intermittent viremic episode with a viral load above detection level but below 200 copies/ml and a return to an undetectable level in a next control).
* Willingness to complete scheduled assessments and participant visits.
* Adequate peripheral vein access to perform leukapheresis
* All female participants of childbearing potential should have a negative pregnancy test. These women and their partner should use double barrier contraception during the study. Females of reproductive potential will need a negative serum or urine pregnancy test at screening. They are defined as those who have not reached menopause or been post-menopausal for at least 24 consecutive months, who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, specifically hysterectomy, or bilateral oophorectomy or tubal ligation) . NOTE: Acceptable documentation of hysterectomy and bilateral oophorectomy, bilateral salpingectomy, tubal micro-inserts, partner who has undergone vasectomy, and menopause is participant-reported history. All participants must agree not to participate in a conception process (e.g., active attempt to become pregnant, sperm donation, or in vitro fertilization).

Exclusion Criteria:

* Previous or current history of AIDS defining event as defined in category C of the 'Centers for disease control and prevention (CDC)' clinical classification .
* Any acute infection or serious medical illness within 60 days prior to study entry. Participants will be excluded from this study for a serious illness (requiring systemic treatment and/or admission) until the subject either completes therapy or is clinically stable on therapy, in the opinion of the Investigator, for at least 14 days prior to study entry
* History of resistance to antiretroviral drugs, documented by genotyping.
* Active hepatitis B or C virus infection: as defined with a positive serology for either disease with signs of active viral replication?
* Significant risk of HIV transmission during treatment interruption in the opinion of the investigator. This includes evidence for unsafe sexual contacts.
* Current or past history of cardiomyopathy or significant ischemic or cerebrovascular disease.
* History of HIV-related thrombocytopenia.
* Active renal disease (defined as a glomerular filtration rate (calculated by MDRD equation) below 50 ml/min or the presence of HIV associated nephropathy in the past medical history.
* Current or known history of cancer (with the exception of in situ cervix carcinoma or squamous cell carcinoma of the skin) within five years prior to screening.
* Pregnancy and breastfeeding.
* Any condition, including psychiatric and psychological disorders that might interfere with adherence to study requirements or safety of the participant.
* Prior use of any HIV vaccine and/or non-established experimental therapy
* Any of the following laboratory test results at screening: 1. Confirmed hemoglobin <11g/dl for women and <12 g//dl for men 2. Confirmed platelet count < 90,000/μl 3. Confirmed neutrophil count <1200/μl 4. Confirmed AST and/or ALT > 5 x upper limit on normal range (ULN). One retest within 14 days is allowed.
* Receipt of any immune modulator or suppressor within 30 days prior study entry, including, but not limited to drugs such as corticosteroids (with the exception of corticosteroids used for topical use), granulocyte-macrophage colony-stimulating factor, interleukin (IL)-2, IL-7 and IL-15.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Participation in other interventional studies involving investigational drug.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Florence, Dr, Principal Investigator — Institute of Tropical Medicine
Locations (4):
- Belgium (4):
  - Institute of Tropical Medicine, Antwerp
  - Saint-Pierre University Hospital, Brussels
  - Brussels University Hospital, Brussels
  - Ghent University Hospital, Ghent

REFERENCES:
- [Derived] Pannus P, Rutsaert S, De Wit S, Allard SD, Vanham G, Cole B, Nescoi C, Aerts J, De Spiegelaere W, Tsoumanis A, Couttenye MM, Herssens N, De Scheerder MA, Vandekerckhove L, Florence E. Rapid viral rebound after analytical treatment interruption in patients with very small HIV reservoir and minimal on-going viral transcription. J Int AIDS Soc. 2020 Feb;23(2):e25453. doi: 10.1002/jia2.25453. PMID 32107887

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Interruption: The ART treatment in patients with a very low viral reservoir will be interrupted.
  Phase 1: Screening visit for HIV patients. During this visit a blood sample is taken for HIV reservoir analysis. Patients in which the reservoir is below a certain treshold will continue to phase 2 and will have their ART treatment interrupted (treatment interruption period).
Period: Phase 1
Arm/Group | Treatment Interruption
Started | 114
Completed | 16
Not Completed | 98
Not completed — Active hepatitis B or C infection | 1
Not completed — Confirmed neutrophil count <1200/µl | 1
Not completed — Detectable level of HIV DNA or caRNA | 75
Not completed — Subject does not want to participate | 20
Not completed — Lost to Follow-up | 1
Period: Phase 2 - Treatment Interruption
Arm/Group | Treatment Interruption
Started | 16
Completed | 14
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
Groups:
- All Participants (Both Phase 1 and 2): 114 subjects were screened in phase 1. Only those with a low viral reservoir continued to phase 2 (16 subjects).
Arm/Group | All Participants (Both Phase 1 and 2)
Number analyzed (Participants) | 114
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  years
    Phase 1 | 45.5 [38.0 to 52.0]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 43.5 [38.0 to 54.0]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  Participants
    Phase 1: Female | 6
    Phase 1: Male | 108
    Phase 2: number analyzed (Participants) | 16
    Phase 2: Female | 1
    Phase 2: Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  Participants
    Phase 1: Asian | 1
    Phase 1: Black African | 1
    Phase 1: White | 111
    Phase 1: Other: Colombian | 1
    Phase 2: number analyzed (Participants) | 16
    Phase 2: Asian | 0
    Phase 2: Black African | 0
    Phase 2: White | 16
    Phase 2: Other: Colombian | 0
Risk group [Count of Participants; unit: Participants] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  Participants
    Phase 1: Heterosexual contact | 14
    Phase 1: Homo/Bisexual contact | 95
    Phase 1: Transfusion, non-haemophilia related | 1
    Phase 1: Other: unknown | 4
    Phase 2: number analyzed (Participants) | 16
    Phase 2: Heterosexual contact | 3
    Phase 2: Homo/Bisexual contact | 12
    Phase 2: Transfusion, non-haemophilia related | 0
    Phase 2: Other: unknown | 1
Duration of HIV infection (months) [Median (Inter-Quartile Range); unit: months] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  months
    Phase 1 | 70.9 [47.0 to 100.8]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 47.2 [33.1 to 75.3]
Duration of HIV infection (years) [Median (Inter-Quartile Range); unit: years] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  years
    Phase 1 | 5.9 [3.9 to 8.4]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 3.9 [2.8 to 6.3]
Duration of ART (months) [Median (Inter-Quartile Range); unit: months] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  months
    Phase 1 | 51.2 [36.1 to 71.4]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 47.3 [34.4 to 74.0]
Duration of ART (years) [Median (Inter-Quartile Range); unit: years] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  years
    Phase 1 | 4.3 [3.0 to 6.0]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 4.0 [2.9 to 6.2]
Last used ART [Count of Participants; unit: Participants] — II = Integrase Inhibitor; NRTI = Nucleoside Reverse Transcriptase Inhibitor; NNRTI = Non-Nucleoside Reverse Transcriptase Inhibitor; PI = Protease Inhibitor Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  Participants
    Phase 1: II + NRTI | 49
    Phase 1: NNRTI + NRTI | 51
    Phase 1: PI + NRTI | 10
    Phase 1: Other | 4
    Phase 2: number analyzed (Participants) | 16
    Phase 2: II + NRTI | 11
    Phase 2: NNRTI + NRTI | 4
    Phase 2: PI + NRTI | 1
    Phase 2: Other | 0
HIV type [Count of Participants; unit: Participants] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  Participants
    Phase 1: A | 3
    Phase 1: B | 106
    Phase 1: C | 1
    Phase 1: CRF02_AG | 4
    Phase 2: number analyzed (Participants) | 16
    Phase 2: A | 1
    Phase 2: B | 15
    Phase 2: C | 0
    Phase 2: CRF02_AG | 0
Nadir CD4 count [Median (Inter-Quartile Range); unit: cells/µl] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  cells/µl
    Phase 1 | 379.0 [338.0 to 482.0]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 440.5 [342.0 to 500.5]
ALT [Median (Inter-Quartile Range); unit: IU/L] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  IU/L
    Phase 1 | 31.0 [23.0 to 37.0]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 21.5 [17.5 to 29.5]
AST [Median (Inter-Quartile Range); unit: IU/L] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  IU/L
    Phase 1 | 27.0 [21.0 to 31.0]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 21.5 [18.5 to 25.0]
Neutrophil count [Median (Inter-Quartile Range); unit: cells/µL] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  cells/µL
    Phase 1 | 3.1 [2.4 to 4.0]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 2.8 [2.1 to 4.0]
CD4 count [Median (Inter-Quartile Range); unit: cells/µL] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  cells/µL
    Phase 1 | 733.0 [645.0 to 891.0]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 758.0 [679.0 to 845.0]
Creatin [Median (Inter-Quartile Range); unit: mg/dL] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  mg/dL
    Phase 1 | 1.0 [0.9 to 1.1]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 1.0 [0.9 to 1.1]
Hemoglobin [Median (Inter-Quartile Range); unit: g/dL] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  g/dL
    Phase 1 | 15.0 [14.2 to 15.7]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 15.1 [14.5 to 15.9]
HCVAb [Median (Inter-Quartile Range); unit: IU/mL] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  IU/mL
    Phase 1 | 1.0 [0.8 to 1.0]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 1.0 [1.0 to 1.0]
HBsAb [Count of Participants; unit: Participants] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  Participants
    Phase 1: >1000mIU/mL | 32
    Phase 1: Negative | 74
    Phase 1: No result | 8
    Phase 2: number analyzed (Participants) | 16
    Phase 2: >1000mIU/mL | 3
    Phase 2: Negative | 11
    Phase 2: No result | 2
HBcAb [Count of Participants; unit: Participants] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  Participants
    Phase 1: Negative (<0.8 IU/mL) | 61
    Phase 1: Positive (1.0 IU/mL or more) | 38
    Phase 1: Grey Zone (0.8-0.99 IU/mL) | 3
    Phase 1: No result | 12
    Phase 2: number analyzed (Participants) | 16
    Phase 2: Negative (<0.8 IU/mL) | 7
    Phase 2: Positive (1.0 IU/mL or more) | 7
    Phase 2: Grey Zone (0.8-0.99 IU/mL) | 1
    Phase 2: No result | 1
HBsAg [Count of Participants; unit: Participants] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  Participants
    Phase 1: Negative | 100
    Phase 1: Positive | 2
    Phase 1: No results | 12
    Phase 2: number analyzed (Participants) | 16
    Phase 2: Negative | 15
    Phase 2: Positive | 0
    Phase 2: No results | 1
Plasma viral load [Median (Inter-Quartile Range); unit: copies/mL] — A value of 19 means <20 copies/mL (lower limit of detection). Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  copies/mL
    Phase 1 | 19.0 [19.0 to 19.0]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 19.0 [19.0 to 19.0]
Platelets [Median (Inter-Quartile Range); unit: 10^9 cells/L] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  10^9 cells/L
    Phase 1 | 232.0 [199.0 to 260.0]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 239.5 [207.5 to 285.0]
Reservoir CD4 caRNA [Median (Inter-Quartile Range); unit: copies/million CD4+ T-cells] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption). This variable was only tested in those subjects that continued to phase 2 (treatment interruption).
  copies/million CD4+ T-cells
    number analyzed (Participants) | 16
    (all) | 105.5 [64.0 to 280.0]
Ultra-sensitive plasma viral load [Median (Inter-Quartile Range); unit: copies/mL] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption). This variable was only tested in those subjects that continued to phase 2 (treatment interruption).
  copies/mL
    number analyzed (Participants) | 16
    (all) | 0.3 [0.0 to 2.5]
Viral reservoir assay DNA [Median (Inter-Quartile Range); unit: copies/10^6PBMCs] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  copies/10^6PBMCs
    Phase 1 | 107.0 [46.0 to 205.0]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 37.5 [11.5 to 55.5]
Viral reservoir assay RNA [Median (Inter-Quartile Range); unit: copies/10^6PBMCs] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption).
  copies/10^6PBMCs
    Phase 1: number analyzed (Participants) | 16
    Phase 1 | 3.0 [1.0 to 6.0]
    Phase 2: number analyzed (Participants) | 16
    Phase 2 | 2.0 [0.0 to 3.5]
Spontaneous VRA CD4 [Median (Inter-Quartile Range); unit: copies/mL] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption). This variable was only tested in those subjects that continued to phase 2 (treatment interruption).
  copies/mL
    number analyzed (Participants) | 16
    (all) | 1.0 [1.0 to 1.5]
Stimulated VRA CD4 [Median (Inter-Quartile Range); unit: copies/mL] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption). This variable was only tested in those subjects that continued to phase 2 (treatment interruption).
  copies/mL
    number analyzed (Participants) | 16
    (all) | 1.6 [0.5 to 3.0]
Spontaneous VRA PBMC [Median (Inter-Quartile Range); unit: copies/mL] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption). This variable was only tested in those subjects that continued to phase 2 (treatment interruption).
  copies/mL
    number analyzed (Participants) | 16
    (all) | 0.7 [0.0 to 1.0]
Stimulated VRA PBMC [Median (Inter-Quartile Range); unit: copies/mL] — Population: 114 participants were included in phase 1 of the study. 16 of those continued to phase 2 (treatment interruption). This variable was only tested in those subjects that continued to phase 2 (treatment interruption).
  copies/mL
    number analyzed (Participants) | 16
    (all) | 2.2 [0.9 to 3.0]

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Number of Participants With a HIV Plasma Viral Load Below the Lower Limit of Detection 48 Weeks Following Interruption of Antiretroviral Treatment
Description: The number of post treatment controllers (PTC - i.e. patients under ART at baseline that show low peripheral blood proviral DNA and still will show sustained viral suppression at 48 weeks after treatment interruption) will be determined. The assessment will be based on the plasma viral load (expressed in copies/ml) measured two-weekly (or four-weekly after W12) until W48 after treatment interruption. Patients below the lower limit of detection (<50 HIV RNA copies/ml plasma) at 48 weeks after treatment interruption will be considered as PTC.
Time Frame: 48 weeks after treatment interruption
Population: Analysis population contains all subjects enrolled in phase 2 (treatment interruption phase)
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Interruption: The ART treatment in patients with a very low viral reservoir will be interrupted.
  ART interruption
Arm/Group | Treatment Interruption
Number analyzed (Participants) | 16
Participants | 0

2. Secondary Outcome: Number of Patients With and the Severity of Adverse Events That Are Related to the Study Intervention, Graded According to NCI CTCAE Version 4.0
Description: Confirmation of the safety of a treatment interruption strategy in selected patients will be based on the number and intensity of AEs graded according to the NCI Common Terminology Criteria for Adverse Events v4.0 (CTCAE) on a five-point scale (Grade 1 to 5: Mild, Moderate, Severe, Life-threatening and Death).
Time Frame: 23 months
Population: Population analyzed are the subject enrolled in het treatment interruption phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Interruption
Number analyzed (Participants) | 16
Participants
  Fatigue: Mild | 1
  Fatigue: Moderate | 0
  Fatigue: Severe | 0
  Fatigue: Life-threatening | 0
  Fatigue: No AE | 15
  Influenza-like illness: Mild | 1
  Influenza-like illness: Moderate | 0
  Influenza-like illness: Severe | 0
  Influenza-like illness: Life-threatening | 0
  Influenza-like illness: No AE | 15
  Oropharyngeal pain: Mild | 1
  Oropharyngeal pain: Moderate | 0
  Oropharyngeal pain: Severe | 0
  Oropharyngeal pain: Life-threatening | 0
  Oropharyngeal pain: No AE | 15

3. Secondary Outcome: Evaluation of the Reservoir Replenishment Upon Interruption of Antiretroviral Treatment (TI) by Quantifying the Viral Reservoir at Baseline (i.e. Just Before TI) and at Viral Rebound (Total HIV DNA).
Description: Assessment of the viral reservoir magnitude on cryopreserved Peripheral Blood Mononuclear Cells (PBMCs) prior and after treatment interruption by means of Total HIV DNA.
Time Frame: At screening, baseline, week 2, week 4, week 6, week 8 and at 12 weeks after relapse
Population: Population analyzed are the subjects enrolled in phase 2 (treatment interruption).
Measure: Median (Inter-Quartile Range); unit: copies/10^6PBMCs
Groups:
- Phase 2 - Treatment Interruption: The ART treatment in patients with a very low viral reservoir will be interrupted.
Arm/Group | Phase 2 - Treatment Interruption
Number analyzed (Participants) | 16
copies/10^6PBMCs
  Screening | 37.5 [11.5 to 55.5]
  Baseline | 22.5 [4.0 to 53.5]
  Week 2 | 27.5 [11.0 to 69]
  Week 4 | 46.5 [18 to 127]
  Week 6 | 38.0 [22 to 141.5]
  Week 8 | 83.5 [82 to 85]
  Post week 12 | 42.5 [29 to 117]

4. Secondary Outcome: Evaluation of the Reservoir Replenishment Upon Interruption of Antiretroviral Treatment (TI) by Quantifying the Viral Reservoir at Baseline (i.e. Just Before TI) and at Viral Rebound (Unspliced RNA).
Description: Assessment of the viral reservoir magnitude on cryopreserved Peripheral Blood Mononuclear Cells (PBMCs) prior and after treatment interruption by means of unspliced RNA.
Time Frame: At screening, baseline, week 2, week 4, week 6, week 8 and at 12 weeks after relapse
Population: Population analyzed are the subjects enrolled in phase 2 (treatment interruption).
Measure: Median (Inter-Quartile Range); unit: copies/10^6PBMCs
Arm/Group | Phase 2 - Treatment Interruption
Number analyzed (Participants) | 16
copies/10^6PBMCs
  Screening | 2 [0.0 to 3.5]
  Baseline | 7.0 [4.0 to 16.5]
  Week 2 | 7.5 [5.0 to 19.5]
  Week 4 | 23.5 [5.0 to 179]
  Week 6 | 30.5 [10.5 to 177]
  Week 8 | 34.5 [31 to 38]
  Post week 12 | 12 [5 to 15]

5. Secondary Outcome: Assessment of the Kinetics of HIV Viral Load Rebound After Treatment Interruption Based on the Repetitive Plasma Viral Load Measurements.
Description: The kinetics will be on the plasma viral load (expressed in copies/ml) measured two-weekly (or four-weekly after W12) until W48 after treatment interruption. A viral load of 19 means <20 copies/mL (lower limit of detection).
Time Frame: At screening, baseline, week 2, week 4, week 6, week 8, End of Intervention (relapse), 4 weeks after relapse and 12 weeks after relapse
Population: The population analyzed are the subjects enrolled in phase 2 (treatment interruption).
Measure: Median (Inter-Quartile Range); unit: copies/mL
Arm/Group | Phase 2 - Treatment Interruption
Number analyzed (Participants) | 16
copies/mL
  Screening | 19 [19 to 19]
  Baseline | 19 [19 to 19]
  Week 2 | 19 [19 to 55.5]
  Week 4 | 1223 [26 to 40600]
  Week 6 | 4020 [2110 to 21100]
  Week 8 | 3480 [3480 to 3480]
  En of Intervention (moment of relapse) | 28000 [2330 to 44900]
  Post week 4 | 22 [19 to 165]
  Post week 12 | 19 [19 to 26]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the whole study period (from start of treatment interruption until end of follow-up period which was 12 weeks after relapse and treatment restart).
Groups:
- Treatment Interruption: Subjects enrolled in phase 2 (treatment interruption). There was no AE collection during phase 1.
Arm/Group | Treatment Interruption
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 13/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Interruption (N=16)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Influenza-like illness (General disorders) | 4 (4)
Bronchitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4)
Oral herpes (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1)
Vit D deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-07-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT02590354/SAP_000.pdf
  • Study Protocol (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/54/NCT02590354/Prot_001.pdf